CLINICAL TRIAL: NCT07142330
Title: Evaluation of Atherectomy in the Management of Occlusive Lesions of the Common Femoral Arteries (RAFAL)
Brief Title: Evaluation of Atherectomy in the Management of Occlusive Lesions of the Common Femoral Arteries
Acronym: RAFAL
Status: Not yet recruiting | Type: Observational
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Other Study IDs: RAFAL
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Femoral Artery Occlusion; Atheromatous Plaques
MeSH Terms: conditions — Plaque, Atherosclerotic | interventions — Atherectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with scheduled atherectomy
  Interventions: Procedure: Atherectomy

INTERVENTIONS:
Procedure: Atherectomy — Two different techniques : rotational atherectomy or thromboendarterectomy

SUMMARY:
Thromboendarterectomy is the standard technique for the treatment of symptomatic occlusive lesions of the common femoral artery. It consists of surgically controlling the artery and interrupting circulation, opening the vessel and removing the atherosclerotic plaque. However, this technique is associated with healing difficulties, postoperative infections, and debilitating incisional pain. The rise of endovascular therapies, particularly at the coronary level, has led to the emergence of new deocclusion techniques, including rotational atherectomy. This technique relies on the use of an intravascular catheter that reams out the atherosclerotic plaque while re-aspirating the resulting debris. A few studies have examined the use of rotational atherectomy for occlusive lesions of the common femoral arteries, but have not evaluated its results compared to the standard treatment. The aim of this multicenter cohort is to describe the efficacy and safety of rotational atherectomy and the standard treatment, thromboendarterectomy, in symptomatic occlusive lesions affecting the common femoral artery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient over 18 years of age
* Non-emergency
* Claudicating patient with significant de novo calcified stenosis affecting the common femoral artery, technically eligible for revascularization by thromboendarterectomy or rotational atherectomy
* Surgery planned with either technique
* Patient's consent to participate in the study must be obtained,

Exclusion Criteria:

* Patient contraindicated for either technique (for surgical or anesthesiological reasons)
* Patient with asymptomatic lesions of the common femoral artery
* Patient with a history of surgery or angioplasty/stenting of the femoral stump
* Patient with occlusion of the ipsilateral common femoral artery or external iliac artery
* Patient with an indication for additional aortofemoral, iliofemoral, femoral-popliteal, or hamstring bypass
* Patient with severe trophic disorders for which a major amputation is considered immediately in addition to revascularization
* Patient objecting to the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Claudicating patient with significant de novo calcified stenosis affecting the common femoral artery, technically eligible for revascularization by thromboendarterectomy or rotational atherectomy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Local complications | one month
  Local complications are defined as follows: hematoma, active bleeding, local infection, thrombosis, delayed healing, false aneurysm, arteriovenous fistula, and neuropathic pain following surgical trauma.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé de Villeneuve d'Ascq,, Villeneuve-d'Ascq, France